CLINICAL TRIAL: NCT01706744
Title: Can Discharge Via an Intermediate Care Unit Prevent Aggravation of Disease and Loss of Functionality, Without Increasing the Level of Cost? A Controlled Observational Study
Brief Title: Effect of Discharge Via an Intermediate Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009/1697
Record Dates: First submitted 2012-10-11; First posted 2012-10-15 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Patients; Aged
Keywords: Hospital Readmissions; Community Health Services; Preventive Health Services; Norway

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intermediate care unit (Experimental): Follow-up treatment and care in a intermediate care unit after discharge from hospital
  Interventions: Other: Intermediate care unit
- Local health care 1 (Active Comparator): Discharge from hospital to usual care as provided by the local health and social care (Verdal)
  Interventions: Other: Local health care 1
- Local health care 2 (Active Comparator): Discharge from hospital to usual care as provided by the local health and social care (Stjørdal)
  Interventions: Other: Local health care 2

INTERVENTIONS:
Other: Intermediate care unit
  Arms: Intermediate care unit
Other: Local health care 1
  Arms: Local health care 1
Other: Local health care 2
  Arms: Local health care 2

SUMMARY:
The main goal is to investigate the following topics:

1. Can discharge via the Intermediate Care Unit in Stjørdal, compared to direct discharge to Verdal Municipality, be equally effective in preventing aggravation of disease and loss of function for patients over 60 years that have been hospitalized in Levanger hospital?
2. Are the cost by discharge to the Intermediate Care Unit in Stjørdal, when the hospital is not located in the same Municipality, comparable to the cost by direct discharge to the Municipality of Verdal, for patients over 60 years that have been hospitalized in Levanger hospital?
3. Which issues are considered important by patients and health personnel during discharge, arrival and follow up in the Municipality, to ensure an optimal interaction between the involved units.

ELIGIBILITY:
Inclusion Criteria:

Patients 60 years old or older from Stjørdal- or Verdal municipality,

* given consent,
* admitted from their home,
* diagnostics completed and necessary treatment started
* the patient need not less than 3-4 days institutionalization for treatment/rehabilitation/care

Exclusion Criteria:

* Patients with severe dementia
* Patients with severe disease who cannot give consent
* Patients with severe disease with short life expectancy (including severe cancer)

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2010-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Hospital readmission | 30 days
  Acute admission to hospital within 30 days from previous discharge
Use of local health care services | up to 1 year

SECONDARY OUTCOMES:
death | up to 1 year
hospital admission | up to 1 year
functional assessment status | up to 6 months
Health service cost | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Roar Johnsen, PhD, Study Director — Norwegian University of Science and Technology
Locations (4):
- Norway (4):
  - Sykehuset Levanger, Levanger
  - Distriksmedisinsk Senter, Stjørdal
  - Stjørdal Kommune, Stjørdal
  - Verdal kommune, Verdal

REFERENCES:
- [Result] Dahl U, Johnsen R, Saetre R, Steinsbekk A. The influence of an intermediate care hospital on health care utilization among elderly patients--a retrospective comparative cohort study. BMC Health Serv Res. 2015 Feb 1;15:48. doi: 10.1186/s12913-015-0708-4. PMID 25638151
- [Result] Dahl U, Steinsbekk A, Jenssen S, Johnsen R. Hospital discharge of elderly patients to primary health care, with and without an intermediate care hospital - a qualitative study of health professionals' experiences. Int J Integr Care. 2014 Apr 30;14:e011. doi: 10.5334/ijic.1156. eCollection 2014 Apr. PMID 24868194
- [Result] Dahl U, Steinsbekk A, Johnsen R. Effectiveness of an intermediate care hospital on readmissions, mortality, activities of daily living and use of health care services among hospitalized adults aged 60 years and older--a controlled observational study. BMC Health Serv Res. 2015 Aug 28;15:351. doi: 10.1186/s12913-015-1022-x. PMID 26315779